CLINICAL TRIAL: NCT01704469
Title: A Comparison of the Perception of a Needle Injection Pain Between Cancer Patients Receiving Opioid Therapy Versus Opioid-naive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2012-0066
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Cancer Patients
Keywords: Opioid induced hyperalgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The local anesthetic injection group (Experimental)
  Interventions: Procedure: The local anesthetic injection

INTERVENTIONS:
Procedure: The local anesthetic injection

SUMMARY:
Opioid-induced hyperalgesia (OIH) is most broadly defined as a state of nociceptive sensitization caused by exposure to opioids. In humans, the evidence of OIH is strong but conflicting. Previous clinical studies mostly used experimental or non-standardized surgical stimuli to assess OIH. We therefore sought to certify a presence of OIH using a standardized, clinical pain stimuli in cancer patients receiving opioid therapy and opioid-naive patients.

ELIGIBILITY:
Inclusion Criteria:

* age 20-80
* cancer patient
* patient whom receiving opioid treatment, any acute or chronic pain condition amenable to a diagnostic/therapeutic nerve block or neuromodulation,and a regular analgesic regimen.

Exclusion Criteria:

* patient who has any change in opioid or other analgesic medications less than 14 days prior to the scheduled procedure
* an inability to understand English or adequately respond to the relevant questions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Post-injection pain intensity | 1 min after lidocaine anesthetic injection
  The local anesthetic injection before main procedure was performed by one pain physician using a 25-gauge needle and 1 ml of 1% lidocaine to raise a small skin wheel. Before and immediately following the injection, patients were asked to rate injection-specific pain and unpleasantness intensity on a 0 to 10 numerical rating scale (NRS).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea